CLINICAL TRIAL: NCT06255626
Title: A Phase 1/2 Multicenter, Randomized Study of the Safety and Immunogenicity of a Sub-unit Protein CD40.RBDv Bivalent COVID-19 Vaccine, Adjuvanted or Not, as a Booster in Volunteers.
Brief Title: Safety and Immunogenicity of a Sub-unit Protein CD40.RBDv Bivalent COVID-19 Vaccine, Adjuvanted or Not, as a Booster in Volunteers.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Vaccine Research Institute (VRI), France (Unknown); EnnoDc (previously known as LinKinVax) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ANRS0407s - LKV.Cov40; 2023-504594-20-00 (Other: EuCT number)
Record Dates: First submitted 2024-02-08; First posted 2024-02-13 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: COVID-19
Keywords: Vaccine; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — CVnCoV COVID-19 vaccine

STUDY DESIGN:
Masking Description: This is an open label study. Immunological assessors, only, will remain blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 1-CD40.RBDv non adjuvanted or mRNA vaccine (5:1 ratio) (Experimental): Low dose (LD) CD40.RBDv vaccine non adjuvanted or mRNA vaccine (5:1 ratio). If randomized to receive LD CD40.RBDv vaccine non adjuvanted in part 1, the subject will be randomised a second time to receive LD CD40.RBDv vaccine non adjuvanted (1:1) in part 2.
  Following a substancial amendment the randomization to mRNA vaccine has been removed from study design
  Interventions: Drug: CD40.RBDv vaccin (SARS-Cov2 Vaccin)
- 2-CD40.RBDv vaccine adjuvanted or mRNA vaccine (5:1 ratio) (Experimental): LD CD40.RBDv vaccine adjuvanted or mRNA vaccine (5:1 ratio) If randomized to receive LD CD40.RBDv vaccine adjuvanted in part 1, the subject will be randomised a second time to receive LD CD40.RBDv vaccine adjuvanted (1:1) in part 2.
  Following a substancial amendment the randomization to mRNA vaccine has been removed from study design
  Interventions: Drug: CD40.RBDv vaccin (SARS-Cov2 Vaccin)
- 3-High dose (HD) CD40.RBDv vaccine non adjuvanted or mRNA vaccine (5:1 ratio) (Experimental): High dose (HD) CD40.RBDv vaccine non adjuvanted or mRNA vaccine (5:1 ratio) If randomized to receive HD CD40.RBDv vaccine non adjuvanted in part 1, the subject will be randomised a second time to receive HD CD40.RBDv vaccine non adjuvanted (1:1) in part 2.
  Following a substancial amendment the randomization to mRNA vaccine has been removed from study design
  Interventions: Drug: CD40.RBDv vaccin (SARS-Cov2 Vaccin)
- 4-High dose (HD) CD40.RBDv vaccine adjuvanted or mRNA vaccine (Experimental): HD CD40.RBDv vaccine adjuvanted or mRNA vaccine (5:1 ratio) If randomized to receive HD CD40.RBDv vaccine adjuvanted in part 1, the subject will be randomised a second time to receive HD CD40.RBDv vaccine adjuvanted (1:1) in part 2.
  Following a substancial amendment the randomization to mRNA vaccine has been removed from study design
  Interventions: Drug: CD40.RBDv vaccin (SARS-Cov2 Vaccin)

INTERVENTIONS:
Drug: CD40.RBDv vaccin (SARS-Cov2 Vaccin) — 1 or 2 injection(s) of CD40.RBDv vaccine (or mRNA vaccine 1 injection (5:1))
  Other Names: COVID-19 mRNA vaccine

SUMMARY:
The goal of this clinical trial, on healthy volunteers, is to learn more about safety and reactogenicity of the CD40.RBDv vaccine.

The main questions that will be studied are :

* Is the CD40.RBDv (adjuvanted or not) safe ?
* Does the CD40.RBDv (adjuvanted or not) imply an immunologic response ? Participants will receive, depending on their randomization arm, 1 or 2 injections of the CD40.RBDv vaccine or a single injection of approved mRNA vaccine

DETAILED DESCRIPTION:
Phase 1/2a randomized, multicentre trial with four cohorts of two arms in two parts.

Part 1:

Cohort 1: Low dose (LD) CD40.RBDv vaccine non adjuvanted or mRNA vaccine (5:1 ratio)

Cohort 2: LD CD40.RBDv vaccine adjuvanted or mRNA vaccine (5:1 ratio)

Cohort 3: High dose (HD) CD40.RBDv vaccine non adjuvanted or mRNA vaccine (5:1 ratio)

Cohort 4: SC injection of HD CD40.RBDv vaccine adjuvanted or mRNA vaccine (5:1 ratio)

A substancial amendment (January 2025) has removed the randomisation to mRNA vaccine from the study design

Go-criterion for opening enrolment within cohorts are detailed into the protocol.

Part 2 at Month 3 :

Group 1: Volunteers who received mRNA vaccine in Part 1 will not receive any vaccine

Group 2: Volunteers who received a first dose of CD40.RBDv vaccine (adjuvanted or not) in Part 1 but randomized (1:1) to receive no further dose of vaccine in Part 2.

Group 3: Volunteers who received a first dose of CD40.RBDv vaccine (adjuvanted or not) in Part 1 and randomized (1:1) to receive an additional dose of CD40.RBDv vaccine (adjuvanted or not)

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers Age ≥18 and <85
* Able to understand and comply with planned study procedures and sign an informed consent before performance of any study-related screening procedures
* Who has received a primary series of vaccination and ≥ 1 booster(s) of COVID-19 mRNA vaccination(s) with the last boost at least 6 months prior to the inclusion in the study
* Subjects has adequate organ functions, evidenced by normal ALT, AST, and alkaline phosphatase
* Normal haematology lab values
* Negative virology assessment
* Normal Urine testing
* Volunteers must meet the eligibility criteria in the approved package labelling of the active comparator
* For women of childbearing potential: use of an effective contraceptive method and negative pregnancy test. For male participants, use of an effective method of contraception with their partner

Exclusion Criteria:

* Acute febrile infection within the previous 72 hours and/or presenting symptoms suggestive of COVID-19 or SARS CoV 2 infection within the previous 28 days
* Immunosuppressive medications received within last three months before first IMP administration or within 6 months for chemotherapies
* Immunoglobulins within 90 days before first IMP administration
* Blood products within 120 days before first IMP administration
* Any medical condition, such as cancer, that might impair the immune response
* Use of any experimental therapy
* Intent to participate in another study of an investigational research agent within 4 weeks prior to the enrolment visit or until the end of the study
* Currently pregnant or breastfeeding
* History of severe adverse events following vaccine administration
* Any bleeding disorder considered as a contraindication to an intramuscular injection
* A condition that requires active medical intervention or monitoring to avert grave danger to Asthma other than mild, well-controlled asthma.
* Hypertension
* BMI ≥ 40 kg/m2; ≤ 18 kg/m2; or BMI ≥ 35 kg/m2 with 2 or more of the following: age > 45, current smoker, known hyperlipidemia, blood pressure is defined as consistently ≥ 140 mm Hg systolic and ≥ 90 mm Hg diastolic
* Malignancy
* Asplenia
* Seizure disorder
* History of hereditary angioedema acquired angioedema, or idiopathic angioedema
* History of myocarditis, pericarditis, cardiomyopathy, congestive heart failure with permanent sequelae, clinically significant arrhythmia (including arrhythmia requiring medication, treatment, or clinical follow-up
* History of autoimmune disease
* Any medical, occupational, or other condition that, in the judgment of the investigator, would interfere with or serve as a contraindication to protocol adherence
* Psychiatric condition that precludes compliance with the protocol.
* Live attenuated vaccines received within 30 days before first IMP administration or scheduled within 28 days after one of the last injection according to the protocol
* Vaccines that are not live attenuated vaccines and were received within 21 days prior to first IMP administration
* Allergy treatment with antigen injections within 30 days before first IMP administration and until the end of the study

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 215 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants without any grade 3 or 4 biological or clinical solicited local/systemic or unsolicited AEs between D1 and Month 3 after each IMP/vaccine administration and considered to be related or possibly related to IMP administration | Month 3
  These proportions of participants will be described with its 95% two-sided confidence interval.
Neutralization antibodies titers (anti-RBD) against the original strain D614G and the relevant strain circulating at time of the study Month 1 | Month 1
  The primary immunogenecity endpoint is the neutralization antibodies titers (anti -RBD) against the original strain D614G and the relevant strain circulating at time of the study Month 1 after each dose The geometric mean titers (GMTs) with 95% confidence intervals (CIs) will be calculated at baseline and at Month 1 after each dose.

SECONDARY OUTCOMES:
Number of volunteers with solicited local and systemic Adverse Reactions (ARs) | Day 8
  The original verbatim terms used by investigators to identify adverse events in the eCRF will be mapped to preferred terms using the MedDRA dictionary. The adverse events will then be grouped by MedDRA preferred terms into frequency tables according to system organ class. All reported adverse events, as well as adverse events judged by the investigator as at least possibly related to study vaccine, will be summarized according to system organ class and preferred term within system organ class and by interval of study observation. When an adverse event occurs more than once for a participants, the maximal severity and strongest relationship to the vaccine group will be chosen.
Number of volunteers with Adverse Events (AEs) other than solicited adverse events | Day 1 to Months 3 after each dose
  The original verbatim terms used by investigators to identify adverse events in the eCRF will be mapped to preferred terms using the MedDRA dictionary. The adverse events will then be grouped by MedDRA preferred terms into frequency tables according to system organ class. All reported adverse events, as well as adverse events judged by the investigator as at least possibly related to study vaccine, will be summarized according to system organ class and preferred term within system organ class and by interval of study observation. When an adverse event occurs more than once for a participants, the maximal severity and strongest relationship to the vaccine group will be chosen.
Number of volunteers with Serious Adverse Events (SAEs), grade 3 and grade 4 | Day 1 to Months 3 after each dose
  The original verbatim terms used by investigators to identify adverse events in the eCRF will be mapped to preferred terms using the MedDRA dictionary. The adverse events will then be grouped by MedDRA preferred terms into frequency tables according to system organ class. All reported adverse events, as well as adverse events judged by the investigator as at least possibly related to study vaccine, will be summarized according to system organ class and preferred term within system organ class and by interval of study observation. When an adverse event occurs more than once for a participants, the maximal severity and strongest relationship to the vaccine group will be chosen.
Number of volunteers with events leading to discontinuation of the vaccine regimen | Through study completion, an average of 15 months
  The original verbatim terms used by investigators to identify adverse events in the eCRF will be mapped to preferred terms using the MedDRA dictionary. The adverse events will then be grouped by MedDRA preferred terms into frequency tables according to system organ class. All reported adverse events, as well as adverse events judged by the investigator as at least possibly related to study vaccine, will be summarized according to system organ class and preferred term within system organ class and by interval of study observation. When an adverse event occurs more than once for a participants, the maximal severity and strongest relationship to the vaccine group will be chosen.
  Separate summaries will be produced for the following categories:
  * Serious adverse events
  * Adverse events that are possibly or probably related to vaccine
  * Adverse event leading to withdrawal from the study
  * After any vaccination and by vaccination
Seroconversion rate defined by an increase of 4 folds between day1 (baseline before vaccination) and Month 1 in anti-RBD IgG binding titers | Month 1
  • The seroconversion rate defined by an increase of 4 folds between day1 (baseline before vaccination) and Month 1 in anti-RBD IgG binding titers will be described with its 95% two-sided confidence interval.
To assess the cross-neutralization against the most relevant VOCs at the time of the study | Day 1 (before each vaccination) day 8, day 14 and M1 after each vaccination, M3, M6, M12 (ie. 12 months after 1st dose and 9 months after 2nd dose) and M15 (ie. 15 months after 1st dose and 12 months after 2nd dose)
  • To assess the cross-neutralization against the most relevant VOCs, The geometric mean titers (GMTs) with 95% confidence intervals (CIs) will be calculated at each timepoint.
To analyze the correlation between the magnitude of CD4+ specific T cell responses and levels of IgG specific responses | Day 1 (before each vaccination) day 14 after each vaccination, M3, M6, M12 (ie. 12 months after 1st dose and 9 months after 2nd dose) and M15 (ie. 15 months after 1st dose and 12 months after 2nd dose)
  • Correlation between the magnitude of CD4+ specific T cell responses and levels of igG specific responses will be estimated at each timepoint using Pearson or Spearman correlation coefficients, depending on variables distribution.
To characterize the vaccine efficacy by evaluating the number of COVID-19 infections (PCR+) and severity (based on CDC definition) in participants throughout the study follow-up. | Through study completion, an average of 15 months
  • Number of COVID-19 infections (PCR+) and severity (based on CDC definition) throughout the study follow-up.
To evaluate the Cytokine expression patterns of CD4 and CD8 T cells as measured by intracellular cytokine staining assay | Day 1 (before each vaccination) day 14 after each vaccination, M3, M6, M12 (ie. 12 months after 1st dose and 9 months after 2nd dose) and M15 (ie. 15 months after 1st dose and 12 months after 2nd dose)
  • Cytokine expression patterns of CD4 and CD8 T cells, measured by intracellular cytokine staining assay, will be described at each timepoint.
Percentages of T cells producing at least one cytokine after in vitro stimulation | Through study completion, an average of 15 months
  • Recall memory T cell responses, following in vitro restimulation (Epimax technology) on residual samples and depending on the results obtained in the analysis of intracellular cytokine staining assay, will be described.
Concentration (pg/mL) of cytokines produced by stimulated PBMC | Through study completion, an average of 15 months
  • Cytokines produced by stimulated PBMC (Luminex assay) on samples evaluated by Epimax technology will be described.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hopital Henri Mondor, Créteil
  - Hôpital Cochin, Paris

IPD SHARING:
Plan to Share IPD: No